CLINICAL TRIAL: NCT00790426
Title: A Phase II Multi-center, Non-randomized, Open Label Study of TKI258 in FGFR3 Mutated and FGFR3 Wild Type Advanced Urothelial Carcinoma
Brief Title: Phase II Study of TKI258 in Advanced Urothelial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2201; 2008-005870-11 (EudraCT Number); EudraCT 2008-005870-11
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-08

CONDITIONS: Urothelial Cancer
Keywords: Advanced urothelial cancer
MeSH Terms: interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

ARMS (2):
- FGFR3 wild type (Experimental)
  Interventions: Drug: TKI258
- FGFR3 mutant (Experimental)
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258

SUMMARY:
This study will evaluate the efficacy of TKI258 in patients with advanced urothelial cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with transitional cell cancer of the bladder, urethra, ureter, or renal pelvis
* Patients who have archival tumor tissue available for FGFR3 mutational status screening
* Patients with progressive disease
* Patients with measurable disease by RECIST
* Patients previously treated with at least 1 but not more than 3 systemic cytotoxic regimens with at least one of these regimens including at least one of the following: cisplatin, carboplatin, gemcitabine or taxane administered in the perioperative or advanced setting
* Age ≥ 18 years
* WHO Performance Status ≤ 2
* Patients willing and able to take oral medication, follow scheduled visits, treatment plan and laboratory tests
* Patients with signed and witnessed informed consent form
* Patients with adequate organ function

Exclusion Criteria:

* Patients with brain cancer
* Patients with other cancers except for certain skin, cervical & prostate cancers
* Patients who have not recovered from previous cancer treatment
* Patients who have severe and/or uncontrolled medical conditions which could affect participation in the study

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 4 months

SECONDARY OUTCOMES:
Disease control rate | 4 Months
Progression free survival | 4 Months
overall survival | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (8):
  - University of California San Diego - Moores Cancer Center UCSD, La Jolla, California
  - USC/Kenneth Norris Comprehensive Cancer Center Regulatory Contact 3, Los Angeles, California
  - University Chicago Hospital CTKI258A2201, Chicago, Illinois
  - Dana Farber Cancer Institute Dana 1230, Boston, Massachusetts
  - Nevada Cancer Institute Nevada Cancer Institute, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center Memorial Sloan Kettering (2), New York, New York
  - Duke University Medical Center Dept.ofDukeUniversityMedCtr(2), Durham, North Carolina
  - The West Clinic, Memphis, Tennessee
- Novartis Investigative Site, Vienna, Austria
- Canada (2):
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Roma, RM, Italy
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Taiwan (2):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taipei
- United Kingdom (2):
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Southampton

REFERENCES:
- [Derived] Milowsky MI, Dittrich C, Duran I, Jagdev S, Millard FE, Sweeney CJ, Bajorin D, Cerbone L, Quinn DI, Stadler WM, Rosenberg JE, Lochheed M, Sen P, Squires M, Shi M, Sternberg CN. Phase 2 trial of dovitinib in patients with progressive FGFR3-mutated or FGFR3 wild-type advanced urothelial carcinoma. Eur J Cancer. 2014 Dec;50(18):3145-52. doi: 10.1016/j.ejca.2014.10.013. Epub 2014 Oct 30. PMID 25457633
- See also: Results for CTKI258A2201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8383